CLINICAL TRIAL: NCT04845971
Title: Phase II Clinical Trial Evaluating Efficacy and Safety of Oral Immunotherapy With Third Generation Gc Protein Derived Macrophage Activating Factor (GcMAF) in Hospitalized Patients With COVID-19 Pneumonia: the COral-MAF1 Trial
Brief Title: Efficacy and Safety of Oral Immunotherapy With GcMAF in Hospitalized Patients With COVID-19 Pneumonia
Acronym: COral-MAF1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dr. Spadera Lucrezia (Other)
Responsible Party: Sponsor-Investigator, Dr. Spadera Lucrezia, Medical Doctor - Department of Otorhinolaryngology Head and Neck Surgery, Ospedale del Mare
Organization: Ospedale del Mare (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: COral-MAF1 Trial - Version 1.0
Record Dates: First submitted 2020-11-17; First posted 2021-04-15 (Actual); Last update posted 2021-09-08 (Actual); Status verified 2021-04

CONDITIONS: COVID-19 Pneumonia
Keywords: COVID-19; VDBP; GcMAF; colostrum-MAF; oral; food supplement
MeSH Terms: conditions — COVID-19 | interventions — vitamin D-binding protein-macrophage activating factor

STUDY DESIGN:
Intervention Model Description: we reserve the possibility that the study may become parallel
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Adult male and female patients who are hospitalized with COVID-19-induced pneumonia. (Experimental): Eligible patients will be treated with Saisei MAF capsules stronger version, oral administration 2-3 capsules, 3 times per day, 30 minutes before food or in the morning, afternoon and before bed time. The treatment duration will be 21 days. Patients are also provided with nutritional supplementation of Vitamin D3, 10.000 IU per day, monitoring the blood levels of such a vitamin. Efficacy and safety assessments will be performed on Days 0, 7, 14, 21, and 28.
  Interventions: Dietary Supplement: Saisei Maf capsules

INTERVENTIONS:
Dietary Supplement: Saisei Maf capsules — Dietary supplement name: Colostrum MAF, Saisei MAF immunomodulator. Formulation: 148 mg acid-resistant coated capsules, containing 2.3 mg of enzymatically treated bovine colostrum powder and supplementary ingredients The dietary supplement substances: Active ingredien: Enzymatically treated bovine colostrum powder 2.3 mg 1.6 % Supplementary ingredients: Lactase (Derived from yeast) 0,15 mg 0.1 % HPMC (Hydroxypropyl Methylcellulose) acid-resistant capsule 47 mg 31.8 % Microcrystalline cellulose (Derived from pulp) 98,4 mg 66.5 % Dosage for adults: 2 - 10 capsules daily (stronger version 9 capsules daily) Route of administration: oral Contraindication: allergy to dairy product components Precaution: pregnancy and lactation Storage: Can be stored in at + 5 to +25°C, on dry place for up to two years Manufacturer: Saisei Pharma, Osaka, MORIGUCHI city, OKUBO-cho, 3-34-8. Japan
  Other Names: Colostrum MAF, Oral MAF, GcMAF

SUMMARY:
As of August 16, 2020, the severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) has been responsible for more than 21 294 000 infections and about 760 000 deaths worldwide. Accumulating evidence suggests that patients with severe acute COVID-19 pneumonia have a cytokine storm syndrome, or unbalanced hyper-inflammatory response. It is now well known that GcMAF plays a crucial role in immune system regulation as a primary defense against infections. Thus, this multifunctional protein, released into the blood stream, acts as a systemic immune modulator without pro-inflammatory activities. In an animal study, IL-6 level was shown to be dramatically decreased after 21 days of oral administration colostrum MAF. Indeed, data from previous studies and clinical practice have been reported its effectiveness and safety in the treatment of many pathologies such as infectious diseases, some types of cancer, juvenile osteopetrosis, immunological, and neurological diseases. These observations suggest that oral immunotherapy with colostrum-MAF is potentially an effective and well-tolerated treatment for COVID-19 pneumonia. In addition, gastrointestinal involvement is well known in coronavirus infections of animals and humans. The angiotensin-converting enzyme II (ACE2), the entry receptor for SARS-CoV, is highly expressed in proximal and distal enterocytes that are directly exposed to foreign pathogens. It considers the mechanism of SARS-CoV-2 can actively infect and replicate in the gastrointestinal tract. SARS-CoV-2 indirectly damages the digestive system through a chain of inflammatory responses. Delivered topically to the small intestine by an acid-resistant enteric-coated capsule colostrum MAF can directly activate a large number of gut mucosal macrophages for virus control, localizing intestinal inflammation and resolving through driven phagocytic scavenger function. Macrophages in the gastrointestinal mucosa represent the largest pool of tissue macrophages in the body, which besides the local functions are directing the systemic immune response.

DETAILED DESCRIPTION:
Over the last five months, there have been increasing numbers of reports that struggle to understand the pathogenesis of the coronavirus disease 2019 (COVID-19) pandemic. To date, the most commonly investigated hypothesis about the underlying mechanisms of multi-organ failure may be summarized into three main targets: microcirculation dysfunction, overwhelming inflammation and abnormal coagulation. Clinical, radiologic and laboratory findings, as well as preliminary autopsy studies, seem to support this hypothesis. As widely suggested, the systemic cytokine storm could play a key role in the virus-induced tissue damage. Being the knowledge of this issue very scarce, lessons learned from other human pathogenic viruses, with specific reference to human immunodeficiency virus (HIV), could be diriment. Unfortunately, no drug or vaccine has yet been approved to treat human coronaviruses and new interventions based on drugs directly active on the virus itself are likely to require months to years to develop. The main targets of the pharmacologic approaches to COVID-19, especially for the complicated cases, are addressed to modulate the immune system and counteract the overwhelming inflammation. Notably, the mechanisms the investigators have hypothesized about the possible pathogenesis of the cell and tissue damage induced by SARS-CoV-2 seem to provide a common denominator in explaining the effects of most drugs currently in use in the clinical trials: these include antivirals, immunomodulating and/or anti-inflammatory drugs. In particular, based on their antiviral activity, chloroquine and hydroxychloroquine, initially conceived as antimalarial therapeutics, were proposed to treat hospitalized patients with COVID-19, with or without azithromycin, showing promising efficacy in "inhibiting the exacerbation of pneumonia, improving lung imaging findings, promoting a virus negative conversion and shortening the disease course". On the other hand, hydroxychloroquine is the cornerstone of medical therapy in lupus, where it acts as an immunomodulatory without immunosuppressive effects. However, because of the lack of evidence about the efficacy and safety of these drugs, the Italian Medicines Agency on July 17 said it had withdrawn an emergency approval for use of the malaria drug hydroxychloroquine or antivirals as a Covid-19 treatment out of clinical trials. Meanwhile the use of low-molecular-weight heparin for COVID-19 is restricted only to well selected hospitalized patients. Tocilizumab, an IL-6 antagonist, approved for the treatment of rheumatoid arthritis and juvenile idiopathic arthritis, also had initial therapeutic application in critical COVID-19 patients, providing encouraging results. However, the phase III clinical trial (COVACTA) for evaluating tocilizumab in hospitalized patients with severe COVID-19 pneumonia found no difference between tocilizumab versus placebo in intensive care requirements or mortality. The rationale basis for the use of monoclonal antibodies in patients affected by SARS-CoV-2 seems to lie in the so-called systemic cytokine storm. Taking into account the key role of VEGF in enhancing angiogenesis in acute lung injury and ARDS, two trials, evaluating the efficacy of bevacizumab as VEGF antagonist in the treatment of COVID-19 (BEST-PC and BEST-RCT), were also started. In light of pathological findings of pulmonary inflammation with edema and hyaline membrane formation, timely and appropriate use of drugs with understood safety profiles aimed at reducing inflammation, microcirculatory dysfunction, oxidative stress, neoangiogenesis and microthrombotic occlusion, in a targeted way, together with ventilator support, should be considered for the severe patients to prevent and treat ARDS development. It is now well known that GcMAF plays a crucial role in immune system regulation as a primary defense against infections. Based on the aforementioned findings and on documented analogies between SARS-CoV-2 and HIV, the investigators hypothesized that the reduced conversion activity of the Gc protein into the macrophage activating factor (MAF) could have a key role in the dysregulate immune response induced by SARS-CoV-2, just like for HIV infected patients. If this hypothesis is correct, it might help to set a valid strategy of immunotherapy also based on an off-label use of GcMAF in critically ill COVID-19 patients. Serum Gc protein, also known as vitamin D-binding protein (DBP), is a multifunctional protein present in plasma/serum at concentrations of 300-600 mg/L. Stepwise hydrolysis of Gc protein by the inducible membranous β-galactosidase of stimulated B-lymphocytes, and by the Neu-1 sialidase of T-lymphocytes converts it into the active GcMAF.On the contrary, deglycosilation of Gc protein by action of the enzyme alpha-N-acetylgalactosaminidase, named nagalase, secreted from HIV-infected cells leads to lack of macrophage activation and to immunosuppression, as a consequence. It is remarkable that nagalase was demonstrated to be an intrinsic component not only of the envelope glycoproteins gp120 and gp160 of HIV but also of the hemagglutinin (HE) of influenza virus and even produced by neoplastic cells. Indeed, flu-like symptoms with serum nagalase activity similar to the influenza acute state were reported in the early stage of HIV-infection, so that the serum enzyme activity may be detectable at all phases of HIV-infection. Similarly, most COVID-19 patients complained of flu-like symptoms in the early stages of the disease. In addition to the storage and transport of active vitamin D3, GcMAF's effects include macrophage modulation, osteoclast activation, facilitation of neutrophil chemotaxis mediated by C5 derived peptide, superoxide activity, scavenging of circulating G-actin, anti-angiogenetic and anti-tumor properties. Thus, this multifunctional protein, released into the blood stream, acts as a systemic immune modulator without pro-inflammatory activities. This means that any function impairment of Gc-globulin could result in a state of both immunosuppression and uncontrolled inflammation, just like in severe COVID-19. Interestingly, HIV viremia was associated with higher level of biomarkers of inflammation (measured by IL-6), monocyte activation (soluble CD14), and coagulation (D-dimer), leading to increased mortality, as compared with uninfected people. Meanwhile, in COVID-19 patients, in addition to the reduced peripheral lymphocyte counts, mainly CD4+ T and CD8+ T cells, there were found significant high levels of pro-inflammatory cytokines and chemokines. Indeed, GcMAF is not only a simple potent activator for macrophages, but more specifically is able to turn macrophage activity on at the sites of infection/inflammation and then to induce their apoptosis by upregulating caspase activity via the p38 and JNK1/2 pathways when no longer needed. Post-mortem lung observations of patients died of COVID-19 showed the presence of mononuclear cells and macrophages infiltrating air spaces by autopsy. With regards to the anti-oxidant properties, it was assessed that GcMAF promotes the superoxide generating capacity of activated macrophages and the production of nitric oxide (NO). It has been showed that the expression of extracellular superoxide dismutase (EC-SOD) mRNA and protein is cell- and tissue-specific and is prominent in lung, heart, blood vessels, placenta and kidney. In particular, high levels of EC-SOD are present in lung macrophages, alveolar type II cells, fibroblasts, vascular smooth muscle cells, and endothelial cells. EC-SOD limits oxidative stress and preserves NO bioactivity, thus protecting against a number of lung and cardiovascular diseases. Even though only in a minority of cases, COVID-19 may progress to life-threatening complications, including respiratory failure, acute cardiac injury, acute kidney injury, septic shock, disseminated intra-vascular coagulation (DIC), and multi-organ dysfunction. Hypoxemia was found to be associated with interstitial pneumonia and, in 10% to 20% of cases, developed into acute respiratory distress syndrome (ARDS). In this connection, it was documented that ARDS as well as organ dysfunction and septic shock is characterized by actin release which is involved in microvascular impairment. DBP has an additional function in binding monomeric globular (G)-actin with high affinity. Thereby, rapidly removing polymeric actin fibrils from the blood stream, it prevents actin polymers from clogging the micro vessels not unlike fibrinogen/fibrin and consequently platelet aggregation and micro thrombi formation. What the investigators postulated could also explain hypercoagulability with elevated concentrations of D-dimer, fibrin degradation products increase, PT and aPTT prolongation, observed in COVID-19 patients. It has been reported that 71.4% of the non survivors of COVID-19 matched the grade of overt-DIC according to the International Society on Thrombosis and Haemostasis (ISTH) diagnostic criteria for DIC. Murine models deficient in DBP showed lung damage caused by actin polymerization, developing severe acute lung inflammation with vascular leakage, hemorrhage and thickening of the vascular wall after actin injection. Interestingly, the lung was the only organ that showed inflammatory injury after intravenous actin injection. The observed lung inflammation was consistent with alterations to lung microvascular endothelial cells. Indeed, when lung endothelial cells were exposed to DBP-actin complexes in vitro showed enhanced cell death. Reduced levels of DBP were even observed in sepsis and organ dysfunction of trauma patients as well as complete depletion of free DBP in those affected by septic shock. These data could provide support for pathogenic explanations of cellular and tissue damage by SARS-CoV-2 and, at the same time, for the therapeutic use of DBP to bind extracellular actin and counteract microcirculatory alterations. Whereas DBP also binds free fatty acids, it was shown that the administration of GcMAF complexed with oleic acid (OA) via nebulisation or subcutaneous injection led to rapid decrease of blood pressure and increase in splenic blood flow, as a result of a verisimilar synergistic NO release by OA-GcMAF-activated alveolar and splenic macrophages. Severe or critically ill COVID-19 patients developed clinical typical manifestations of shock, even in the absence of overt hypotension. Furthermore, it was found that GcMAF can inhibit the angiogenesis induced by pro-inflammatory prostaglandin E1, which serves roles in the promotion of VEGF expression. A key role of VEGF in acute lung injury and ARDS was confirmed. Reflecting the fact that clinical features and severity of symptoms vary widely between and within each COVID-19 patient, with older males more likely to be affected and in a more severe manner, the investigators sought to relate it with some special feature of DBP. Several studies showed that the polymorphisms of DBP were associated with susceptibility or resistance to disease states including chronic obstructive pulmonary disease. Moreover, whereas androgens were not found to have any effect on circulating levels of DBP, exposure to high levels of estrogens increased them by up to 50%, suggesting a potential protective role of estrogens against COVID-19. On the other hand, in relation to vitamin D status, advanced age was recognized as one of the major risk factors for vitamin D deficiency. Animal-based studies also demonstrated that deficiencies in both dietary protein- and energy-intake decreased the concentration of DBP in the circulation. These data seem to be in line with the growing evidence that vitamin D supplementation could reduce the risk of COVID-19 infections and deaths. The present trial aims to assess the efficacy and safety of immunotherapy with oral MAF plus standard-of-care therapy in hospitalized adult patients with COVID-19- induced pneumonia.

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥ 18 years of age);
* signed informed consent by any patient capable of giving consent, or, when the patient is not capable of giving consent, by his or her legal/authorized representative or according to local guidelines;
* patients clinically diagnosed with SARS-CoV-2 virus by PCR or by other approved diagnostic methodology;
* hospitalized with COVID-19-induced pneumonia evidenced by chest x-ray or CT scan with pulmonary infiltrates;
* patients having a PAO2/FIO2 ratio > 250 mmHg;
* well-selected patients having a PAO2/FIO2 ratio ≤ 250 mmHg that, in the investigator's judgment, doesn't preclude the patient's safe participation in and completion of the study;
* patients being able to swallow.

Exclusion Criteria:

* Proportion of hospitalized patients requiring invasive mechanical ventilation at the time of hospital admission (patients requiring non-invasive mechanical ventilation are eligible);
* uncontrolled systemic infection (other than COVID-19);
* hypersensitivity to the active substance or to any of the excipients of the experimental drug, including known allergy to dairy product;
* any serious medical condition or abnormality of clinical laboratory tests;
* in the opinion of the investigator, progression to death is imminent and highly likely within the next 24 hours, irrespective of the provision of treatments;
* current participation in any other interventional investigational trials;
* pregnant or breastfeeding woman;
* concurrent malignancy requiring chemotherapy;
* renal insufficiency;
* all types of disability.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2020-11-05 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
the rate of transfer to the intensive care unit (ICU) | 28 days or until discharge
  the proportion of hospitalized patients requiring intensive care management because of worsening respiratory function (PaO2/FiO2 ratio <150 mmHg) and/or development of multi-organ dysfunction and/or other clinical conditions needing invasive mechanical ventilation Given that 26% of patients required intensive care unit treatment, the purpose of this trial is to achieve a reduction of at least 50% of this value with an overall rate of transfer to the ICU of 13%.

SECONDARY OUTCOMES:
Changes from baseline to subsequent timepoints (when available) in terms of percentage of lung involvement (lung consolidation, ground glass opacities and disease free). | 28 days or until discharge
  CT visual quantitative evaluation will be based on summing up the acute lung inflammatory lesions involving each lobe, which was scored as 0 (0%), 1 (1-25%), 2 (26-50%), 3 (51-75%), or 4 (76-100%), respectively. In particular, an early reduction from 85% to 50% in imaging progression on chest CT at day 7 will be evaluated, as a surrogate endpoint
duration of hospital stay | 28 days or until discharge
  expressed in days
days on non-invasive ventilation | 28 days or until discharge
  expressed in days
time to reduction of FiO2 > 25% | 28 days or until discharge
  expressed in days
days with use of supplemental O2 | 28 days or until discharge
  expressed in days
discharge rate at day 28 | 28 days or until discharge
  expressed in days
clinical evolution | 28 days or until discharge
  proportion of patients with COVID-19 symptoms worsening.
time to resolution of fever | 28 days or until discharge
  time to resolution of fever (for at least 48 hours) in absence of antipyretics, or discharge, whichever is sooner in the 4-week period after study treatment. Resolution of fever is defined as body temperature: ≤36.6°C (axilla) or ≤37.2 °C (oral), or ≤37.8 °C (rectal or tympanic). Fever is defined as defined as body temperature > 37.4°C [axilla], or > 38.0 °C [oral], or >38.4°C [rectal or tympanic];
progression of respiratory failure | 28 days or until discharge
  progression of respiratory failure as evaluated by the PaO2/FiO2 ratio
implementation of supplemental oxygen | 28 days or until discharge
  proportion of patients requiring implementation of supplemental oxygen during the 28-day period
changes from baseline in white blood cell count (WBC) | 28 days or until discharge
  changes from baseline in white blood cell count (WBC)
changes in hemoglobin level | 28 days or until discharge
  changes from baseline in hemoglobin
changes in platelet count | 28 days or until discharge
  changes from baseline in platelets
changes in CRP levels | 28 days or until discharge
  changes from baseline in CRP
changes in ESR value | 28 days or until discharge
  changes from baseline in ESR
changes in LDH levels | 28 days or until discharge
  changes from baseline in LDH
changes in procalcitonin value | 28 days or until discharge
  changes from baseline in procalcitonin
changes in IL-6 levels | 28 days or until discharge
  changes from baseline in IL-6
changes in TNF-α levels | 28 days or until discharge
  changes from baseline in TNF-α
changes in D-dimer | 28 days or until discharge
  changes from baseline in D-dimer
changes in fibrinogen levels | 28 days or until discharge
  changes from baseline in fibrinogen
MAF precursor activity of serum Gc protein | 28 days or until discharge
  changes from baseline in MAF precursor activity of serum Gc protein as marker for response to treatment
serum nagalase activity | 28 days or until discharge
  changes from baseline in serum nagalase activity, as marker for response to treatment;
viral loads detected in nasopharyngeal swabs | 28 days or until discharge
  kinetic changes of viral loads detected in nasopharyngeal swabs
Serious Adverse Events (SAE) and Adverse Drug Reaction (ADR) (expected and unexpected) | 28 days or until discharge
  number of Serious Adverse Events (SAE) and Adverse Drug Reaction (ADR) (expected and unexpected)
patient compliance with treatment. | 28 days or until discharge
  proportion of patients

CONTACTS AND LOCATIONS:
Overall Officials: LUCREZIA SPADERA, MD, Principal Investigator — Department of Otorhinolaryngology Head and neck Surgery - Ospedale del Mare Hospital, naples, Italy
Locations (1):
- Ospedale del Mare Hospital, Naples, Italy

IPD SHARING:
Plan to Share IPD: Undecided
This is a multicenter trial. However, we reserve the possibility of enrolling further COVID-19 Hospital Units that are interested in participating in the trial, in order to get the correct sample size as needed for the study.Thus, if needed, we'll share IPD with the involved research centers.

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2021-02-23): https://cdn.clinicaltrials.gov/large-docs/71/NCT04845971/Prot_SAP_ICF_001.pdf